CLINICAL TRIAL: NCT00622219
Title: Mentored Clinical Career Award in Adolescent Substance Abuse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Sharon Levy, Assistant Professor of Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: K23DA019570 (NIH)
Record Dates: First submitted 2008-02-11; First posted 2008-02-22 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Substance-Related Disorders
Keywords: Alcohol abuse; Drug abuse
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug Testing (Experimental): Adolescents in the experimental condition will receive all of the services offered by the Adolescent Substance Abuse Program (including individual meetings, parent and adolescent group meetings, psychopharmacology as indicated)and will be enrolled in a random drug testing program (with an average of 12 requests for testing over a 12 week period).
  Interventions: Other: Randomized Drug Testing Trial
- Control (No Intervention): Adolescents randomized to the control condition will receive all of the services offered by the Adolescent Substance Abuse Program (including individual meetings, parent and adolescent group meetings, psychopharmacology as indicated) but will not be called for drug tests.

INTERVENTIONS:
Other: Randomized Drug Testing Trial — Adolescents in the experimental condition will receive all of the services offered by the Adolescent Substance Abuse Program (including individual meetings, parent and adolescent group meetings, psychopharmacology as indicated)and will be enrolled in a random drug testing program (with an average of 12 requests for testing over a 12 week period).
  Arms: Drug Testing

SUMMARY:
The goal of this project is to determine the barriers to, and risks and benefits of random laboratory drug testing for adolescents with identified drug or alcohol problems.

DETAILED DESCRIPTION:
Use of drugs and alcohol is associated with a variety of health care problems, making settings where adolescents receive routine medical care ideal for implementation of routine screening and early intervention. However, little research has been conducted on the efficacy of interventions for adolescent primary care patients who are using drugs or alcohol. Urine drug testing can be used for a variety of indications, including school or work based population surveillance, verification of history, or monitoring of individuals who are in treatment for a drug-use disorder. This study will focus exclusively on the therapeutic use of urine drug testing. Drug testing can be a useful therapeutic adjuvant for patients with drug-use disorders in a variety of settings.

This study will investigate the use of random laboratory drug testing as a therapeutic intervention for teens with drug problem use, abuse or dependence. We have 5 objectives:

1. To develop a standardized protocol for random urine drug testing, produce a manual and training protocol, and refine the protocol in preparation for a future efficacy trial.
2. To estimate the cost of a random drug-testing program.
3. To determine the factors that are associated with willingness to be tested, and barriers to enrolling adolescents in laboratory drug testing programs.
4. To perform an initial, small-scale experimental trial of the random drug testing protocol. The purpose of this trial is to estimate the effect size of the intervention and will be used in calculating the sample size for a future stage 1b trial.
5. To determine the potential risks to adolescents who participate in a random drug testing program, including possible breach of confidentiality, greater conflict between the parent and child, more difficulty with communication between clinician and patient, increased use of drugs not detected by routine urine screens (i.e. inhalants), and increased use of strategies and products known to defeat drug tests.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents ages 12-21
* Participants must have use of alcohol, cannabis, or another substance on at least 2 occasions in the 30 days preceding their initial assessment or 6 or more times in the past 90 days
* Participants must have health insurance or be willing to pay for the laboratory costs associated with drug testing.
* Participants must provide informed assent and, for those under 18, parental consent.

Exclusion Criteria:

* Participants who require immediate hospitalization or immediate referral to residential substance abuse treatment
* Participants who cannot understand or read English at a 6th grade reading level
* Participants who are enrolled in the ASAP buprenorphine program
* Participants who report previous use of inhalants or any other substance that is not easily detected with urine drug testing

Ages: 12 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2008-03; Primary Completion 2013-08-31 (Actual); Study Completion 2013-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage days abstinent from any substance use during the past 90 days, as measured by self-report via a Time Line Follow Back calendar (TLFB). | 90 days

SECONDARY OUTCOMES:
Adolescent willingness to participate a in drug testing program. | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Levy, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States

REFERENCES:
- [Background] Levy S, Harris SK, Sherritt L, Angulo M, Knight JR. Drug testing of adolescents in ambulatory medicine: physician practices and knowledge. Arch Pediatr Adolesc Med. 2006 Feb;160(2):146-50. doi: 10.1001/archpedi.160.2.146. PMID 16461869
- [Background] Levy S, Harris SK, Sherritt L, Angulo M, Knight JR. Drug testing of adolescents in general medical clinics, in school and at home: physician attitudes and practices. J Adolesc Health. 2006 Apr;38(4):336-42. doi: 10.1016/j.jadohealth.2005.11.023. PMID 16549293
- See also: web site of the Center for Adolescent Substance Abuse Research at Children's Hospital Boston — http://www.ceasar.org